CLINICAL TRIAL: NCT00196625
Title: Study on Safety and Efficacy of Salvage Therapy With Amprenavir, Lopinavir and Ritonavir 200 Mg/d or 400 Mg/d in HIV-Infected Patients in Virological Failure.ANRS 104 PUZZLE 1
Brief Title: Salvage Therapy With Amprenavir, Lopinavir and Ritonavir in HIV-Infected Patients in Virological Failure.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 104 PUZZLE1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: HIV infections; Salvage therapy; Amprenavir; Lopinavir; Ritonavir
MeSH Terms: conditions — HIV Infections | interventions — amprenavir; Pharmaceutical Preparations; Ritonavir

INTERVENTIONS:
Drug: Amprenavir (drug)
Drug: ABT-378/r (drug)
Drug: Ritonavir (drug)

SUMMARY:
HIV infected patients are treated with highly active antiretroviral therapy (HAART). Side effects and the great number of pills reduces adherence to the treatment, and induces therapeutic failure. In order to maintain efficacy of HAART, new combination is evaluated. The aim of the study is to compare the antiviral efficacy of this salvage therapy combining lopinavir and amprenavir with 200 mg/d or 400 mg/d ritonavir, together with nucleoside reverse transcriptase inhibitors, over a 26-week period in HIV-infected patients in whom multiple antiretroviral regimens had failed.

DETAILED DESCRIPTION:
HIV infected patients are treated with highly active antiretroviral therapy (HAART). Side effects and the great number of pills reduces adherence to the treatment, and induces therapeutic failure. In order to maintain efficacy of HAART, new combination is evaluated. The aim of the study is to compare the antiviral efficacy of this salvage therapy combining lopinavir and amprenavir with 200 mg/d or 400 mg/d ritonavir, together with nucleoside reverse transcriptase inhibitors (NRTI), over a 26-week period in HIV-infected patients in whom multiple antiretroviral regimens had failed. 100 patients with CD4 cell count below 300/mm3 and plasma HIV RNA over 30,000 copies/ml are to be included in four groups: amprenavir, lopinavir, NRTI, with ritonavir 200 mg.d or not (patients previously treated by additional ritonavir 200 or 400 mg/d).

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* CD4 cell count below 300/mm3
* Plasma HIV RNA over 30,000 copies/ml
* Previously treated with 2 protease inhibitors and 1 non nucleoside analogue (except amprenavir, lopinavir)
* Written informed consent

Exclusion Criteria:

* Biological abnormalities
* Pregnancy
* Alcool abuse
* History of pancreatitis, hepatic failure
* Acute HIV related infection
* Chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2000-11; Study Completion 2002-02

PRIMARY OUTCOMES:
Mean change of VIH RNA between week 0 and week 26

SECONDARY OUTCOMES:
Disease progression
CD4 cell count
Safety
Pharmacokinetics
Genotypic resistance

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Raguin, MD, Principal Investigator — Service des Maladies Infectieuses et Tropicales, Hôpital Saint-Antoine, Paris, France; Genevieve Chene, MD, PhD, Study Director — INSERM U593, Bordeaux, France

REFERENCES:
- [Result] Raguin G, Chene G, Morand-Joubert L, Taburet AM, Droz C, Le Tiec C, Clavel F, Girard PM; Puzzle 1 Study Group. Salvage therapy with amprenavir, lopinavir and ritonavir 200 mg/d or 400 mg/d in HIV-infected patients in virological failure. Antivir Ther. 2004 Aug;9(4):615-25. PMID 15456093
- [Result] Taburet AM, Raguin G, Le Tiec C, Droz C, Barrail A, Vincent I, Morand-Joubert L, Chene G, Clavel F, Girard PM. Interactions between amprenavir and the lopinavir-ritonavir combination in heavily pretreated patients infected with human immunodeficiency virus. Clin Pharmacol Ther. 2004 Apr;75(4):310-23. doi: 10.1016/j.clpt.2003.12.013. PMID 15060509